CLINICAL TRIAL: NCT04949880
Title: The Efficacy and Safety Study for Endovascular Treatment of Symptomatic Intracranial Atherosclerotic Stenosis Using Neurovascular Drug-Eluting Balloon Dilatation Catheter: A Prospective Multicentre Single-arm Trial
Brief Title: A Single-Arm Trial of Neurovascular Drug-Eluting Balloon Dilatation Catheter Treating Symptomatic Intracranial Atherosclerotic Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYLOX34202105
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Intracranial Atherosclerosis
MeSH Terms: conditions — Intracranial Arteriosclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental): Neurovascular Drug-Eluting Balloon Dilatation Catheter
  Interventions: Device: Neurovascular Drug-Eluting Balloon Dilatation Catheter

INTERVENTIONS:
Device: Neurovascular Drug-Eluting Balloon Dilatation Catheter — The neurovascular drug-eluting balloon dilatation catheter consists of a tip, a drug-coated balloon, markers, a catheter and a catheter hub. The main component of the drug coating is sirolimus, and the coating is evenly distributed on the effective length surface of the balloon.

SUMMARY:
This is a trial designed to test the efficacy and safety of the Neurovascular Drug-Eluting Balloon Dilatation Catheter.

DETAILED DESCRIPTION:
This is a prospective multicentre single-arm trial conducted by 11 centers in mainland China. Approximately 132 subjects with symptomatic intracranial atherosclerotic stenosis receive endovascular treatment using the neurovascular drug-eluting balloon dilatation catheter designed by Zylox.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years, any gender;
* Subject has symptomatic intracranial atherosclerotic stenosis that the degree of the artery stenosis is between 70% and 99% diagnosed by intracranial angiography;
* The target stenotic artery locates in Internal Carotid Artery (intracranial segment), Middle Cerebral Artery (M1, M2), Basilar Artery, Vertebral Artery (intracranial segment);
* Intracranial artery stenosis requiring interventional treatment is a single lesion;
* Subject has at least two atherosclerosis risk factors including history or present hypertension, diabetes, hyperlipidemia, smoking, age>45;
* modified Rankin Scale(mRS) score≤2 before enrollment;
* Subject or guardian is able to understand the purpose of study, agree to provide follow-up data and has provided written informed consent.

Exclusion Criteria:

* History of acute ischemic stroke within 2 weeks;
* History of intracranial hemorrhage (including intraparenchymal hemorrhage, subarachnoid hemorrhage, subdural hemorrhage and epidural hemorrhage) within 3 months;
* Hypertension uncontrolled by medicine (Systolic pressure≥180 mmHg or diastolic pressure≥110 mmHg continuously);
* Combined with the intracranial tumor, aneurysm or intracranial arteriovenous malformation;
* The length of intracranial artery stenosis >10mm and extremely angulated >90°, which indicated by angiography;
* History of stent intervention within the target lesion;
* Allergic to heparin, sirolimus (i.e. rapamycin), contrast agents, aspirin, clopidogrel, anesthetics;
* History of gastrointestinal hemorrhage within 6 months before signing the informed consent form, which is unable to receive antiplatelet therapy;
* Platelet (PLT)<90*10^9/L;
* Creatinine>250 umol/L;
* International Normalized Ratio (INR)>1.5;
* Female subject who is pregnant or breast-feeding, or who has a pregnancy plan within 12 months;
* Expected life <12 months;
* Unable to cooperate with or tolerate the interventional surgery;
* Subject who has participated in other drug or device clinical trials or hasn't reached the primary end point;
* Angiography indicates intracranial artery stenosis caused by arterial dissection, arteritis, and thrombosis;
* Angiography indicates the vascular path is tortuous, the experimental device is difficult to reach the target position or be retracted;
* Other circumstances judged by researchers that are not suitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Restenosis rate of the target lesion | 180+60 days
  Subjects receive Digital Subtraction Angiography (DSA) / Computed Tomography Angiography (CTA) examination in 180 days to analyze whether the degree of stenosis is greater than or equal to 50%, if so, the target lesion restenosis happens.

SECONDARY OUTCOMES:
Average stenosis degree of the target lesion | 180+60 days
  Subjects receive DSA / CTA examination in 180 days.
Success rate of device | Intraoperation
  After receiving DSA examination, success rate of device is defined as experimental device-neurovascular drug-eluting balloon dilatation catheter advanced on position successfully, balloon retracted smoothly after expanded, without balloon rupture and balloon catheter break, etc.
Success rate of surgery | Intraoperation
  After receiving DSA examination, success rate of surgery is defined as the final residual stenosis degree of target lesion<50% and modified thrombolysis in cerebral infarction score (mTICI) 2b/3, whether or not other additional treatments are applied.

OTHER OUTCOMES:
Incidence of device deficiency | within 180+60 days
  Device deficiency is the unreasonable risk that may endanger human health and life safety in the normal use of medical devices during clinical trials, such as labeling errors, quality problems, malfunctions, etc.
Incidence of stroke events | 7 days or at discharge / 30±7 days / 180+60 days
  Stroke events include hemorrhagic or ischemic stroke, transient cerebral ischemia.
Rate of death | 7 days or at discharge / 30±7 days / 180+60 days
  Subjects who died from any cause would be counted.
The rate of AE | within 180+60 days
  The definition of AE (Adverse Event) refers to ISO 14155.
The rate of SAE | within 180+60 days
  The definition of SAE (Serious Adverse Event) refers to ISO 14155.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital; Liqun Jiao, Principal Investigator — Xuanwu Hospital, Beijing
Locations (11):
- China (11):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Cangzhou Central hospital, Cangzhou, Hebei
  - Wuhan Hospital of Traditional Chinese and Western Medicine, Wuhan, Hubei
  - General Hospital of Northen Theater Command, Shenyang, Liaoning
  - Linyi People's Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Changhai Hospital of Shanghai, Shanghai